CLINICAL TRIAL: NCT00480610
Title: Clinical Study on Tacrolimus Ointment Over the Long-term. "CONTROL Study - Adults"
Brief Title: Treatment and Control of Atopic Dermatitis With 0.1% Tacrolimus Ointment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FG-506-06-40
Record Dates: First submitted 2007-05-30; First posted 2007-05-31 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-09

CONDITIONS: Dermatitis, Atopic
Keywords: Dermatitis, atopic; Tacrolimus; Adult; treatment outcomes
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Tacrolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: tacrolimus ointment
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo ointment

INTERVENTIONS:
Drug: tacrolimus ointment — Topical application
  Other Names: Protopic®
  Arms: 1
Drug: Placebo ointment — Topical application
  Arms: 2

SUMMARY:
Long-term tacrolimus ointment based regimen comprising of up to 6 weeks of initial twice daily treatment and subsequent twice weekly prophylactic application can effectively treat active lesions of atopic dermatitis and prevent delay & reduce flares

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient of any ethnic group
* Patient was at least 16 years old and suffered from mild to severe atopic dermatitis (Rajka/Langeland score of at least 3)

Exclusion Criteria:

* Patient had a genetic epidermal barrier defect such as Netherton's syndrome or generalised erythroderma
* Patient had a clinically significant skin infection on the affected (and to be treated) area

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2004-04; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Number of exacerbations of atopic dermatitis requiring intervention. | 12 months

SECONDARY OUTCOMES:
Time to first exacerbation requiring intervention; exacerbation treatment days, periods and time to first exacerbation; physician and patient assessment of affected area, treatment response; quality of life; global response | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Principal Investigator — Klinik und Poliklinik für Dermatologie und Allergologie, Ludwig-Maximilians Universität
Locations (22):
- Innsbruck, Austria
- Belgium (2):
  - Brussels
  - Edegem
- Prague, Czechia
- Aarjus, Denmark
- Helsinki, Finland
- France (2):
  - Paris
  - Saint-Etienne
- Germany (4):
  - Bonn
  - Dresden
  - Düsseldorf
  - München
- Italy (2):
  - Modena
  - Roma
- Netherlands (2):
  - Amsterdam
  - Utrecht
- Almada, Portugal
- Spain (2):
  - Barcelona
  - Madrid
- Geneva, Switzerland
- United Kingdom (2):
  - Cardiff
  - Southhampton

REFERENCES:
- [Background] Wollenberg A, Reitamo S, Girolomoni G, Lahfa M, Ruzicka T, Healy E, Giannetti A, Bieber T, Vyas J, Deleuran M; European Tacrolimus Ointment Study Group. Proactive treatment of atopic dermatitis in adults with 0.1% tacrolimus ointment. Allergy. 2008 Jul;63(7):742-50. PMID 18592619
- [Background] Wollenberg A, Sidhu MK, Odeyemi I, Dorsch B, Koehne-Volland R, Schaff M, Ehlken B, Berger K. Economic evaluation of maintenance treatment with tacrolimus 0.1% ointment in adults with moderate to severe atopic dermatitis. Br J Dermatol. 2008 Dec;159(6):1322-30. doi: 10.1111/j.1365-2133.2008.08807.x. Epub 2008 Sep 6. PMID 18782316